CLINICAL TRIAL: NCT05073068
Title: Timed Exercise to Acutely Improve Energy and Substrate Metabolism at Night in Men and Women With Prediabetes
Brief Title: Acute Timed Exercise and 24h Metabolism
Acronym: TIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: NL78628.068.21
Record Dates: First submitted 2021-08-25; First posted 2021-10-11 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2024-12

CONDITIONS: Type 2 Diabetes; Overweight and Obesity
Keywords: Day-night rhythm; Metabolism; Metabolic flexibility; Exercise; Glycogen
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participants will receive a code so that the person in charge with the data quality check and the data analyses will be blinded to the interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- AM exercise (Experimental)
  Interventions: Behavioral: Timing of exercise
- PM exercise (Experimental)
  Interventions: Behavioral: Timing of exercise
- Control (Active Comparator)
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Timing of exercise — An acute exercise bout of cycling performed in the morning at 9 AM or at 5 PM
  Arms: AM exercise; PM exercise
Behavioral: Control — No exercise
  Arms: Control

SUMMARY:
The primary objective of this randomized controlled cross-over study is to investigate if an acute, glycogen lowering exercise bout performed either in the morning or late afternoon differentially affects the respiratory exchange ratio at night in men and women with prediabetes. For this purpose, participants will stay in a respiration chamber and will be subjected to either an exercise bout in the morning or late afternoon.

DETAILED DESCRIPTION:
Appropriate timing of lifestyle interventions may facilitate healthy rhythmicity in metabolism and optimize the effectiveness of such interventions in improving metabolic health. In this context, exercise is well-known to improve (skeletal muscle) energy metabolism and is an established intervention to improve muscle insulin sensitivity and to counter the development of type 2 diabetes (T2D). In addition, exercise may also have beneficial effects on the immune response that is known to impact on insulin sensitivity and overall metabolic health. In this study it is hypothesized that exercise performed at different times of the day exerts a differential effect on 24h metabolism in people at risk for developing T2D. To test this, a randomized controlled cross-over study is conducted in which participants are subjected to either an exercise in the morning or late afternoon while staying in the respiration chamber. Main outcome is substrate utilization during the night as measured with the respiration chamber, but 24-hrs blood draws will also be performed to examine effect of exercise on circulating metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Healthy (determined by dependent physician)
* Man or post-menopausal woman
* Age between 50 - 75 years
* BMI ≥ 25 kg/m2
* Pre-diabetes based on meeting at least one of the following criteria: impaired glucose tolerance defined as plasma glucose values ≥ 7.8 mmol/l and ≤ 11.1 mmol/l 120 minutes after glucose drink consumption during oral glucose tolerance test in screening, impaired fasting glucose defined as fasting plasma glucose ≥ 6.1 mmol/l and ≤ 6.9 mmol/l, insulin resistance defined as a glucose clearance rate ≤ 360 mL/kg/min as determined using OGIS120, HbA1c of 5.7-6.4%
* Regular sleeping habits (7 - 9h of daily sleep)
* Stable diet and weight: No weight gain or loss > 3kg in the last three months

Exclusion Criteria:

* Not meeting all inclusion criteria
* Fasting plasma glucose
* ≥ 7.0 mmol/L
* Hemoglobin < 7.8 mmol/L
* Previously diagnosed with type 2 diabetes
* Uncontrolled hypertension
* In case of an abnormal electrocardiogram at rest: this will be discussed with the responsible medical doctor
* Subjects who do not want to be informed about unexpected medical findings during the screening /study, or do not wish that their physician is informed
* Any contra-indication to the Equivital telemetric pill
* Hypomotility disorders of the gastro-intestinal tract
* Extreme early bird or extreme night person (score ≤30 or ≥70 on morning-eveningness questionnaire self assessment)
* Heavily varying sleep-wake rhythm
* Night shift work during last 3 months
* Travel across > 1 time zone in the last 3 months
* Frequent engagement in programmed exercise as judged by the investigator
* Significant food allergies/intolerance (seriously hampering study meals)
* Participation in another biomedical study within 1 month before the first study visit
* Using > 400mg caffeine daily (more than 4 cups of coffee or energy drinks)
* Smoking
* Any acute condition, exacerbation of chronic condition, or medical history that would in the investigator's opinion interfere with the study
* Antecubital veins that present tremendous difficulty in obtaining frequent blood draws (e.g. too small)

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2024-11-21 (Actual); Study Completion 2024-11-21 (Actual)

PRIMARY OUTCOMES:
Nocturnal respiratory exchange ratio | 35 hours respiration chamber stay per intervention arm
  Relative carbohydrate/fat oxidation during the night

SECONDARY OUTCOMES:
24 hour energy and substrate metabolism determined using oxygen and carbondioxide levels as measured with whole-chamber respirometry | 35 hours respiration chamber stay per intervention arm
Immune cell phenotypes determined using blood samples obtained during the interventions | 35 hours respiration chamber stay per intervention arm
Blood glucose levels following the exercise intervention measured continuously using a continuous glucose monitor device | 7 days post the exercise intervention

OTHER OUTCOMES:
Diurnal variation in circulating glucoregulatory hormones (e.g. insulin) analysed in blood samples obtained throughout the day | 35 hours respiration chamber stay per intervention arm
Feet sensitivity based on score on a neuropathy questionnaire | Baseline visit
Diurnal variation in metabolite levels (e.g. glucose, free fatty acids) analysed in blood samples obtained throughout the day | 35 hours respiration chamber stay per intervention arm
Diurnal variation in core body temperature using a core temperature pill that measures 24hrs | 35 hours respiration chamber stay per intervention arm
Feet sensitivity based on a clinical foot assessment | Baseline visit

CONTACTS AND LOCATIONS:
Overall Officials: Joris Hoeks, Dr, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No
Participant data will only discussed with other researcher on group level. We are not interested in individual participant data